CLINICAL TRIAL: NCT00774813
Title: Phase II Study Using Nexalin Therapy for the Treatment of Depressive Symptoms Associated With Mild to Moderate Depression Episodes
Brief Title: Nexalin Therapy for the Treatment of Depressive Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kalaco Scientific, Inc. (Industry)
Responsible Party: Evgeny Kruptisky, MD, PhD, Leningrad Regional Center of Addiction
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPMS-7003
Record Dates: First submitted 2008-07-03; First posted 2008-10-17 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Depression
Keywords: Depression; Mild; Moderate; Anxiety; Kalaco Scientific, Inc.
MeSH Terms: conditions — Depression; Lymphoma, Follicular; Anxiety Disorders | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Nexalin 1.3mA device + placebo antidepressant
  Interventions: Device: Nexalin 1.3mA Device
- B (Active Comparator): Nexalin 15mA device + placebo antidepressant
  Interventions: Device: Nexalin 15mA device
- C (Placebo Comparator): Placebo device + SSRI (Citalopram or similar)
  Interventions: Drug: placebo device and Citalopram

INTERVENTIONS:
Device: Nexalin 1.3mA Device — * 3 treatment cycles (cycle is 5 daily treatments, followed by 2 days off)
  * Daily receipt of placebo antidepressant
  Other Names: Nexalin Device
  Arms: A
Device: Nexalin 15mA device — * 3 treatment cycles (cycle is 5 daily treatments, followed by 2 days off)
  * Daily receipt of a placebo antidepressant
  Other Names: Nexalin Device
  Arms: B
Drug: placebo device and Citalopram — * 3 treatment cycles (cycle is 5 daily treatments, followed by 2 days off)
  * Daily receipt of a a SSRI (Citalopram or similar)
  Other Names: Nexalin Device
  Arms: C

SUMMARY:
The primary objectives of this Phase II study are to demonstrate the safety of Nexalin Therapy and to investigate the efficacy of Nexalin Therapy.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, multi-center trial has 3 different treatment arms.

Study Tools:

* Hamilton Depression Rating Scale (HAM-D21)
* Clinical Global Impressions (CGI)
* Montgomery-Asberg Depression Rating Scale (MADRS)
* Beck's Depression Inventory
* Hamilton Anxiety Rating Scale (HAM-A)
* Hospital Anxiety and Depression Scale (HADS)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mild to moderate depression episode, based on the HAM-D21 Rating Scale (10-13 = mild; 14-17 = mild to moderate)
* Diagnosed with mild to moderate depression episode based on ICD-10 Diagnostic Guidelines
* Is willing and able to spend 4 weeks as a hospital inpatient
* Is willing and able to return to the clinic during follow-up period

Exclusion Criteria:

* A HAM-D21 Rating Scale of <10 or >17
* Diagnosed outside of mild to moderate depression episode range based on the ICD-10 Diagnostic Guidelines
* Unable to complete wash-out interval without taking antidepressants or psychotropic medications
* Is pregnant or may be pregnant
* Sensitivity to electrodes and/or their conductive gels or adhesives
* Break in skin integrity at the areas of electrode placement
* Currently taking immune suppressing drugs or suspected use of narcotics
* Presence of any implanted electronic devices, cardiac stimulator, or pacemaker
* History of brain injury, including seizures, epilepsy, stroke, tumor of central nervous system, or hydrocephalus
* History of heart attacks, congestive heart failure, or uncontrolled hypertension
* History of schizophrenia or manic-depressive syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAM-D21) | Screening; Baseline; Treatments 5, 10, & 15; Follow-up Weeks 2, 4, 8, & 12

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) | Screening; Baseline; Treatments 5, 10, & 15; Follow-up Weeks 2, 4, 8, & 12
Montgomery-Asberg Depression Rating Scale (MADRS) | Screening; Baseline; Treatments 5, 10, & 15; Follow-up Weeks 2, 4, 8, & 12
Beck's Depression Inventory | Screening; Baseline; Treatments 5, 10, & 15; Follow-up Weeks 2, 4, 8, & 12
Hamilton Anxiety Rating Scale (HAM-A) | Screening; Baseline; Treatments 5, 10, & 15; Follow-up Weeks 2, 4, 8, & 12
Hospital Anxiety and Depression Scale (HADS) | Screening; Baseline; Treatments 5, 10, & 15; Follow-up Weeks 2, 4, 8, & 12
Medication Usage Log | Every visit
Adverse Event Log | Every visit

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Kruptisky, MD, PhD, Principal Investigator — Leningrad Regional Center of Addiction
Locations (2):
- Russia (2):
  - Leningrad Regional Center of Addiction, Saint Petersburg, Vsevolozhsky District
  - St. Petersburg City Center of Neuroses, Saint Petersburg